CLINICAL TRIAL: NCT06095479
Title: Ultrasound Liver Fat Quantification on Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips (China) Investment CO., LTD (Industry)
Collaborators: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ICBE-S-000403
Record Dates: First submitted 2023-10-12; First posted 2023-10-23 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-05

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- undergo standard abdominal ultrasound imaging and MRI-PDFF (Experimental): Study-related procedures will consist of one investigational exam conducted with the Philips EPIQ Ultrasound System with investigational LFQ software and a standard MRI-PDFF examination.
  All imaging procedures (investigational LFQ ultrasound exam and MRI-PDFF exam) must be completed within an 8-week window (+ 5 days).
  Interventions: Device: 2D ultrasound scan and MRI examination

INTERVENTIONS:
Device: 2D ultrasound scan and MRI examination — All subjects will undergo a 2D ultrasound scan and MRI examination.

SUMMARY:
This prospective study aims to recruit pediatric patients with confirmed or suspected non-alcoholic fatty liver disease (NAFLD) / non-alcoholic steatosis hepatitis (NASH) and who are eligible for standard ultrasound and MRI examinations. All subjects will undergo a 2D ultrasound scan and MRI examination. Approximately 108 subjects will be enrolled, targeting at 90 completing the study.

DETAILED DESCRIPTION:
This prospective study aims to recruit pediatric patients with confirmed or suspected non-alcoholic fatty liver disease (NAFLD) / non-alcoholic steatosis hepatitis (NASH) and who are eligible for standard ultrasound and MRI examinations. All subjects will undergo a 2D ultrasound scan and MRI examination. Approximately 108 subjects will be enrolled, targeting at 90 completing the study.

To assess the correlation between the quantitative ultrasound biomarkers, i.e., HRIQ, AttenQ and ElastQ, and the liver fat content percentage measured by MRI proton density fat fraction (MRI-PDFF) on pediatric patients, in order to evaluate the technical feasibility of using HRIQ, AttenQ and ElastQ to quantify liver fat content for pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects at age of 6-18 years old (≥6 & <18) who are able to provide assent to participate and have a parent/legal guardian who is able to provide informed consent for the subject to participate.
* Subject must be eligible for a standard abdominal ultrasound examination and standard non-contrast MRI examination.
* In addition, at least one of the following criteria must also be met:

  * Overweight or obese (BMI-for-age ≥ 85th percentile).
  * Diagnosed with Type II diabetes per standard clinical guidelines.
  * Diagnosed with hypercholesterolemia per standard clinical guidelines.
  * Diagnosed with or clinically suspected of having NAFLD/NASH based on previous medical record, medical imaging, liver biopsy, and/or laboratory testing.

Exclusion Criteria:

* Evidence of hepatotoxicity in the clinical judgment of the investigator.
* History of chronic liver disease (e.g., viral hepatitis, cholestatic hepatitis, or autoimmune liver disease).
* Use of drugs associated with hepatic steatosis1: amiodarone, aethotrexate, nucleoside reverse transcriptase inhibitors (didanosine, stavudine), valproic acid, dexamethasone, tamoxifen, 5-FU-based adjuvant chemotherapy, apo-B inhibitors (mipomersen, lomitapide), tetracycline exceeding 2 g/day and acetylsalicylic acid exceeding 150 mg/kg.

Note: patients taking tetracycline (≤ 2 g/day), acetylsalicylic acid (≤150 mg/kg) are allowed to be enrolled.

* Subjects with hepatic lesions that cannot be excluded from the imaging field during ultrasound LFQ data acquisition.
* Subjects anticipated or planned to undergo any therapeutic intervention during enrollment period that, at discretion of the Investigator, may affect liver fat content (e.g., bariatric surgery, chemotherapy).
* History of previous liver surgery or hepatic implants that, at the discretion of the Investigator, may adversely impact ultrasound or MRI image quality or the subject's eligibility to undergo ultrasound or MRI.
* Subjects with unstable clinical status, late stages of a given disease, or unpredictable clinical course of a given disease.
* Subjects with evidence of COVID-19 or with the substantial risk of COVID-19 infection.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2023-11-18 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Rate of HRIQ, AttenQ and ElastQ, and the liver fat content percentage measured by MRI | up to 28 months
  To assess the correlation between the quantitative ultrasound biomarkers, i.e., HRIQ, AttenQ and ElastQ, and the liver fat content percentage measured by MRI proton density fat fraction (MRI-PDFF) on pediatric patients, in order to evaluate the technical feasibility of using HRIQ, AttenQ and ElastQ to quantify liver fat content for pediatric patients.

SECONDARY OUTCOMES:
The concentration of robustness of the investigational LFQ software in the clinical settings | up to 28 months
  To assess the inter-operator variability on the same day and the data acquisition failure rate (i.e., the percentage of the subjects whose image quality is unacceptable due to technical limitations) of these quantitative ultrasound biomarkers, in order to evaluate the robustness of the investigational LFQ software in the clinical settings.

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhua Hospital affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, China, China

IPD SHARING:
Plan to Share IPD: No